CLINICAL TRIAL: NCT03499548
Title: The INSPiRe Programme: A Feasibility and Acceptability Study of Intensive Suicide Prevention Therapy in Prison
Brief Title: The INSPiRe Programme: Developing an Intensive Suicide Prevention Therapy for Suicidal Prisoners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Jessica Killilea, University of Manchester, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 238927
Record Dates: First submitted 2018-03-19; First posted 2018-04-17 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Suicide
Keywords: Intensive; Cognitive Behavioral Therapy; Male prisoners
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): 10 hours of intensive CBT for suicide will be delivered to male prisoners who are having thoughts of ending their lives. This will be delivered in 2 hours sessions, 5 times across 2 weeks.
  Interventions: Other: INSPiRe Programme

INTERVENTIONS:
Other: INSPiRe Programme — Intensive CBT for suicide

SUMMARY:
This study aims to assess the acceptability and feasibility of a short-term, intensive Cognitive Behavioural Therapy (CBT) delivered to male prisoners who have thoughts of ending their lives.

DETAILED DESCRIPTION:
10 hours of an adapted CBT therapy for suicide will be delivered across 2 weeks in 5 2 hour sessions to male prisoners. They will initially be assessed on several measures of mood, social support and suicidality. They will then undergo therapy. Following this they will be asked to re-completed the initial measures and a post-therapy interview to ascertain their thoughts on their experience of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 21 years old.
* Has been managed under the Assessment, Care in Custody, and Teamwork (ACCT) system within the last 1 month (including current ACCT review).
* Sufficient English language proficiency, as judged by the researcher, in order to complete psychometric questionnaires (i.e. adequate reading comprehension) and engage in intensive CBT programme (i.e. adequate verbal communication).
* Adult is able to provide informed consent as established during baseline clinical interview (BPS, 2006; MCA, 2005).
* Currently residing in HM Prison (and expected to remain there for at least six weeks; determined through staff and prisoner report).

Exclusion Criteria:

* A primary organic disorder (indicated by prison medical staff report or records).
* Any current risk behaviour which would compromise the safety of others, as identified by prison staff.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants will be recruited from a prison site that houses males.
Enrollment: 13 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
The Client Satisfaction Questionnaire (CSQ-8) | 20 minutes
  A measure of participant satisfaction with therapy
Therapist Session Summary | 5 minutes
  Measuring levels of adherence and engagement
Discharge summary sheet | 15 minutes
  Capturing individuals' adherence to the programme or discharge from it
Therapist Rating Form | 20 minutes
  Giving an overall picture of each individual's engagement and progress during the study.
Post-intervention interview | 1 hour
  Qualitative interview to explore the participant's experience of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pratt, Principal Investigator — University of Manchester; Yvonne Awenat, Study Chair — University of Manchester; Charlotte Lennox, Study Chair — University of Manchester
Locations (1):
- HMP Risley, Warrington, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No